CLINICAL TRIAL: NCT06512012
Title: Technology-Assisted Yoga and Exercise on Chemotherapy-Induced Peripheral Neuropathy and Pain in Children With Leukemia
Brief Title: Technology-Assisted Yoga and Exercise on Neuropathy and Pain in Children With Leukemia
Acronym: yogaCIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/26-75
Record Dates: First submitted 2023-08-28; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Leukemia; Children With Cancer; Yoga Therapy; Excercise; Neuropathy;Peripheral; Pain
Keywords: yoga, excercise, pain, neuropathy, children, leukemia
MeSH Terms: conditions — Leukemia; Neuritis; Pain | interventions — Yoga; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga and exercise group (Experimental): Before starting yoga, "How are you feeling today?" will be asked to child. The yoga session will be individualized according to how the child feels. The content of the yoga sessions will progress in the form of warm-up exercises - breathing work - yoga postures (asana) - meditation - and progressive muscle relaxation exercises. Yoga sessions will be scheduled for 30 minutes. Yoga sessions and progressive muscle relaxation exercises will be held online once a week for eight weeks, then every two weeks for four months.
  Interventions: Behavioral: yoga and exercise
- control group (No Intervention): no yoga or excersize intervention.

INTERVENTIONS:
Behavioral: yoga and exercise — Technology-Assisted Yoga and Exercise Intervention during 6 months
  Arms: Yoga and exercise group

SUMMARY:
The study was planned to examine the effects of technology-supported yoga and exercise on chemotherapy-induced peripheral neuropathy and pain in children aged 5-18 years with leukemia.

DETAILED DESCRIPTION:
The research will be carried out in Marmara University Istanbul Pendik Training and Research Hospital Pediatric Hematology and Oncology Service, and Dokuz Eylul University Pediatric Hematology and Oncology Service. It was planned to include all patients who were selected by the block randomization method, and who met the sampling criteria, in the study. Yoga will be given to the intervention group online. The control group will not be interfered with. Follow-up will be made using data collection tools after taking the study, 3 months later, and 6 months later.

Before starting yoga, "How are you feeling today?" will be asked to child. The yoga session will be individualized according to how the child feels. The content of the yoga sessions will progress in the form of warm-up exercises - breathing work - yoga postures (asana) - meditation - and progressive muscle relaxation exercises. Yoga sessions will be scheduled for 30 minutes. Yoga sessions and progressive muscle relaxation exercises will be held online once a week for eight weeks, then every two weeks for four months.

All yoga sessions will pay attention to the following items:

* Yoga sessions will be stretched according to the child's energy level and comfort.
* If the child expresses that he or she is not feeling well, that yoga session can only consist of breathing exercises and cooling poses.
* The child will be encouraged to express that he/she feels tired when he/she is tired.
* He will be told to move slowly to ensure safety when entering and exiting balance poses.
* The child will be asked what part of his/her body he/she feels while in the pose and where the tension occurs. This will ensure that the child remains safe in the pose.
* If a member of the family wishes to participate while the child is doing yoga, their participation will be supported.
* Movements will be continued by protecting the area with the catheter so that any catheter in the child's body is not bent, twisted, or dislodged.
* Back bending poses with high intensity will not be done.

ELIGIBILITY:
Inclusion Criteria:

* Age range of the child is between 6-18,
* Diagnosed with acute lymphoblastic leukemia,
* Induction (Steroid and Vincristine) treatment,
* Being on an inpatient or outpatient treatment,
* Newly diagnosed or on induction therapy for less than one month,
* child agreeing to participate in the study voluntarily,
* Parent agreeing to participate in the study voluntarily,
* No relapse,
* Obtaining the consent form from the child and the parent,
* The child does not have a physical or psychological deficit,
* The child's yoga and exercise have an electronic device and internet to participate in the intervention.

Exclusion Criteria:

* The patient's relapse or terminal period,
* The child and family are not willing to participate in the study,
* The child has a cognitive, physical, and psychological deficits,
* The child's illiteracy.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Pediatric Modified Total Neuropathy Scale and Total Neuropathy Score-Pediatric Vincristine (TNS-PV) for peripheral neuropathy | during 6 months (at the beginning of the study, 3rd month and 6th month)
  Pediatric Modified Total Neuropathy Scale and Total Neuropathy Score-Pediatric Vincristine (TNS-PV) assessment tools will be used. They determine Chemotherapy-induced Peripheral Neuropathy and its severity in children receiving cancer treatment. Each category is scored between 0-4. The highest 32 points are obtained from the scale. The higher the score, the worse the neuropathy. TNS-PV is based on adding constipation and hoarseness to the Pediatric Modified Total Neuropathy Scale.
Adolescent Pediatric Pain Scale for pain | during 6 months (at the beginning of the study, 3rd month and 6th month)
  Adolescent Pediatric Pain Scale: This scale consists of three independent parts;
  1. body outline diagram where the child/adolescent can mark the location of the pain
     *Assessment: The child can mark the anterior and posterior sides-upper extremity, lower extremity, head, neck, abdomen, chest, shoulder, back… so that the location and number of the pain area is evaluated
  2. 10 cm long, where the pain can mark the severity as "no pain, mild pain, moderate pain, very pain and worst pain possible" word chart scale
     * Evaluation: With a scale of 0-10 cm, the pain is evaluated by the child between 0-10 and the pain is defined as "no pain, mild pain, moderate pain, very pain".
     and defines its intensity by choosing one of the "worst pain possible"
  3. word list under 4 dimensions (sensory, emotional, evaluative, time) to indicate the nature of pain.

SECONDARY OUTCOMES:
Pediatric Symptom Screening Scale for chemotherapy related symptoms | during 6 months (at the beginning of the study, 3rd month and 6th month)
  Pediatric Symptom Screening Scale: It was developed to evaluate the symptoms experienced by children. The scale consists of a total of 15 items and is Likert type.
  The scale score ranges from 0 to 60. The overall score increases as the symptoms worsen.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, Assoc. Prof., Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)